CLINICAL TRIAL: NCT05296616
Title: The Effect of Mindfulness-Based Stress Reduction Intervention on Sleep Quality, Stress Level and Heart Rate Variability of University Students
Brief Title: Sleep Quality, Stress Level and Heart Rate Variability of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Merve BAT TONKUŞ, Lecturer, İstanbul Yeni Yüzyıl Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/03-835
Record Dates: First submitted 2022-03-17; First posted 2022-03-25 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Sleep Quality; Stress Level; Heart Rate Variability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSQSLHRV (Experimental): The group in which the mindfulness-based stress reduction intervention will be implemented.
  Interventions: Behavioral: Mindfulness Based Stress Reduction Intervention
- Control (No Intervention): The group to which mindfulness-based stress reduction intervention will not be applied

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Intervention — Mindfulness Based Stress Reduction intervention is a manualized course that includes meditation, relaxing movement, and breathing. A certified MBSR instructor will teach the courses in a group-based format for 90 minute sessions, once per week for eight weeks.
  Arms: MSQSLHRV

SUMMARY:
Purpose: This study aims to determine the impact of mindfulness-based stress reduction programs on sleep quality, stress level and heart rate variability of university students Design: The study was planned as an experimental study with a randomized control group, using pre-test, post-test and follow-up test.

Hypotheses:

H1: The sleep quality level scores of the students in the intervention group participating in the mindfulness-based stress reduction initiative will increase compared to the students in the control group. H2: Students in the intervention group participating in the mindfulness-based stress reduction initiative will decrease their stress level level scores compared to the students in the control group. H3: The heart rate variability of the students in the intervention group participating in the mindfulness-based stress reduction initiative will be higher than the students in the control group.

H4: The sleep quality level posttest and follow-up scores of the students in the intervention group participating in the mindfulness-based stress reduction initiative will increase compared to their pretest scores. H5: The stress level posttest and follow-up scores of the students in the intervention group participating in the mindfulness-based stress reduction initiative will increase according to their pretest scores. H6: The heart rate variability level posttest and follow-up scores of the students in the intervention group participating in the mindfulness-based stress reduction initiative will increase according to their pretest scores.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of the relevant faculty,
* No barriers to accessing technology for participation in the online program,
* No visual or hearing impairment

Exclusion Criteria:

* Not being a student of the relevant faculty,
* Having barriers to accessing technology for participation in the online program,
* Having visual or hearing impairment

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-18 (Estimated); Primary Completion 2022-11-18 (Estimated); Study Completion 2023-01-18 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality Level | for 8 months
  The Pittsburgh Sleep Quality Index: The 18 items scored are divided into 7 component scores. Some ingredients consist of a single substance, while others are obtained by combining several substances. Each item is assessed on a scale between 0-3. These components are; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction. The sum of these seven component scores gives the overall index score. Your total score is between 0-21. A high total score indicates poor sleep quality. The index does not indicate the presence or prevalence of sleep disorders.

SECONDARY OUTCOMES:
Stress Level | for 8 months
  Perceived Stress Scale is a scale consisting of 14 questions. Participants in the study evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)." The Perceived Stress Scale includes 7 (items 4.5.6.7.9.10. and 13.) reverse scored statements. Total scale scores range from 0 to 56. An increase in the total score indicates an increase in the perceived stress level of the individual.
Heart Rate Variability | for 8 months
  CorSense HRV monitors were purchased from the Elite HRV company for use in the study. Readings will be collected through the Elite HRV app designed for mobile devices.
  RMSSD and LF/HF data will be received for each reading from the application. According to the Elite HRV website, the platform includes RMSSD calculations for the R-R range recorded by industry standards and defines 0.04-0.15 Hz waves as LF and 0.15-0.40 Hz waves as HF.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Bat Tonkus, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No